CLINICAL TRIAL: NCT00823173
Title: An Open Label Exploratory Study to Assess the Safety, Tolerability and Clinical Activity of Topically Applied ESBA105 in Patients With Acute Anterior Uveitis
Brief Title: Exploratory Study on Topical ESBA105 in Acute Anterior Uveitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ESBATech AG (Industry)
Responsible Party: Sushanta Mallick, Head Clinical Trial Management, ESBATech AG
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESBA105CRD04
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2011-05-26 (Estimated); Status verified 2010-09

CONDITIONS: Anterior Uveitis
Keywords: Uveitis; TNF-alpha; Topical; ESBA105; scFv antibody fragment; ocular inflammation
MeSH Terms: conditions — Uveitis, Anterior; Uveitis | interventions — ESBA105

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Topical ESBA105 (Experimental): ESBA105 applied as eye drops
  Interventions: Biological: ESBA105

INTERVENTIONS:
Biological: ESBA105 — ESBA105 eye drops (10mg/mL), initially applied in hourly dosing intervals, followed by later dose tapering (prolongation of dosing intervals)

SUMMARY:
The purpose of this study is to determine whether ESBA105, a topically applied TNF-alpha inhibitor, is safe and clinically active when applied to the eye of patients suffering from acute anterior uveitis

DETAILED DESCRIPTION:
Acute anterior uveitis (AAU) is a common, recurrent disease characterized by inflammation of the iris and ciliary body. Though usually effectively treated by topical corticosteroids, novel treatment modalities are required to overcome the limitations and adverse effect problems associated with the use of corticosteroids. TNF-alpha has been recognized as a central disease mediator in AAU, as shown by preclinical models and clinical data with systemically applied TNF-alpha inhibitors.

ESBA105 is a topically applied TNF-alpha inhibitor that is characterized by efficient penetration into the eye resulting in high intraocular drug levels. A recently completed Phase I trial confirmed that safety and tolerability of topical ESBA105 in healthy individuals is excellent and systemic exposure is low.

In this pilot trial, the safety, local tolerability and clinical activity of topical ESBA105 in the treatment of patients with acute anterior uveitis shall be explored.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent.
* Patients with the typical presentation of HLA-B27 positive AAU (unilateral, painful anterior uveitis of sudden onset).
* 2+ anterior chamber cells according to the SUN Working Group criteria, as assessed by slit lamp biomicroscopy.
* Start of the typical first symptoms of the current attack, defined as the point in time when the patient felt the first sensation of the attack, within the last 72 hours before initiation of treatment with the study medication.
* Negative pregnancy test for females of childbearing potential (pre menopausal, <2 years post-menopausal, not surgically sterile).
* Patients with a negative QuantiFERON TB Gold test result.
* Patients who currently have no clinically apparent symptoms of an HLA B27 associated acute extraocular disorder requiring systemic immunosuppressive therapy.
* Patients who are willing and able to cooperate with study requirements.

Exclusion Criteria:

* IOP elevation requiring therapy.
* Uncontrolled diabetes mellitus and diabetic retinopathy.
* Patients with a single eye or a pinhole Snellen visual acuity 20/200 or worse in the non study eye.
* Patients with 1+ or less anterior chamber cells.
* Patients with 3+ or 4+ anterior chamber cells or hypopyon.
* Patients in whom the time of the beginning of the current attack can not be determined.
* Patients exhibiting corneal ulceration or a history of recurrent herpetic keratitis or clinical evidence of herpetic dermatitis.
* Patients currently treated with topical corticosteroids.
* Patients treated with systemic immunosuppressive therapy within the last 2 months.
* Patients treated with a systemically administered TNF-alpha inhibitor within the last 2 months.
* Pregnant or breast-feeding women or women of childbearing potential, who with their partners refuse to use 2 reliable methods of contraception (including 1 barrier method) during the study.
* Male patients with a female partner who could become pregnant and who refuse, with their partner, to use 2 reliable methods of contraception (including 1 barrier method) during the study.
* Patients whose clinical presentation is suggestive for an active bacterial, viral or fungal infection anywhere in the body.
* Patients with history of recurrent infections, or a clinical presentation suggestive of a chronic infection requiring antimicrobial therapy (e.g. syphilis) including active episodes of serious viral infections by, e.g. herpes simplex, herpes zoster, cytomegalic or hepatitis viruses or clinical signs of fungal infections, such as histoplasmosis, aspergillosis or coccidiomycosis.
* Patients presenting with higher intraocular pressure in the uveitic eye than in the contralateral eye.
* Patients with known carrier status of human immunodeficiency virus, hepatitis B or hepatitis C.
* Patients with a history of demyelinating disease (multiple sclerosis) or optic neuritis.
* Patients with positive or unclear QuantiFERON TB Gold test result or history of high risk exposure to Mycobacterium tuberculosis.
* Patients with known coexisting malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Changes in the level of intraocular inflammation (anterior chamber cell count according to SUN Working group criteria) | 28 Days

SECONDARY OUTCOMES:
Nature and incidence of adverse events, physical and ophthalmological findings and laboratory test results | 28 Days
Systemic exposure to study drug | 28 Days
Changes in disease severity as assessed by visual analogue scale (VAS) | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Zierhut, MD, Study Chair — Universitäts-Augenklinik Tübingen
Locations (3):
- Germany (3):
  - Universitäts-Augenklinik, Tübingen, Baden-Würtemberg
  - Uveitis-Zentrum Franziskus Hospital, Münster, North Rhine-Westphalia
  - Charité Humboldt University, Berlin, State of Berlin